CLINICAL TRIAL: NCT01038648
Title: Does the DPP4 Inhibitor Sitagliptin Have a Role in Preventing Type 2 Diabetes- A Randomised Controlled Study.
Brief Title: Sitagliptin in Prevention of Type 2 Diabetes Mellitus
Acronym: SITAGLIPTIN
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Responsible Party: A. Ramachandran / Chairman / Managing Director / President, IDRF & ARH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SITAGLIPTIN-003 IDRF
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes
Keywords: Sitagliptin; Type 2 diabetes; Prevention of type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Advice life style at baseline only
  Interventions: Other: life style modification at base line
- sitagliptin arm : 2 (Active Comparator): 100mg/day sitagliptin
  advice on life style modification at baseline only
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — 100mg/day
  Arms: sitagliptin arm : 2
Other: life style modification at base line — Advice on physical activity, diet and drug adherence.
  Arms: 1

SUMMARY:
The hypothesis is, in subjects with persistent impaired glucose tolerance(IGT) , sitagliptin will decrease the conversion rate to diabetes as compared to a placebo in three years.

DETAILED DESCRIPTION:
The DPP-4 inhibitor Sitagliptin may be a suitable preventive agent in subjects with IGT or IFG on account of observed functional improvements in islet cell function and potential protective effect on beta cell mass.

Objectives of the study

1. Primary objectives :

   - To test whether the DPP4 inhibitor Sitagliptin is effective in preventing conversion of IGT to diabetes when compared with a placebo.
2. Secondary objectives:

   * To assess rates of reversal from IGT to Normal Glucose Tolerance (NGT) in IGT patients administered Sitagliptin
   * To assess the effect of Sitagliptin on measure of beta cell function and insulin resistance in patients with IGT.

Study design

Double blind placebo controlled, parallel group study - three years follow up .

Subjects with IGT in the age group of 30-55 years (n=900) will be identified by screening with a standard OGTT. Selected subjects will be randomized to the control arm using placebo and the two study arms using Sitagliptin. At baseline all group will receive a standard advice on lifestyle modification. The dose of sitagliptin will be 100 mg/d. The subjects will be reviewed at 6 monthly intervals and repeat OGTT will be done annually.

Proforma containing details of anthropometry, occupation, physical activity, diet habits, details of medications, regularity of treatment and biochemical investigations will be filled up at each interview.

Investigations:

Initial Screening

1. Demographic data
2. Height, weight, waist and hip measurements.
3. Details of family history of diabetes, hypertension and cardiovascular diseases.
4. History of any other major illness.
5. History of blood pressure and measurements.
6. Details of education and occupation.
7. Diet habits will be analyzed by dietician.
8. Details of physical activity will be assessed by a questionnaire.

Laboratory investigations:

1. Initial OGTT
2. Plasma glucose and HbA1c.
3. Lipid profile
4. Liver function tests
5. Serum amylase and serum lipase
6. Plasma insulin
7. 12 lead ECG.

Review analysis:

1. Review will be done with all clinical and biochemical assessment annually.
2. Evaluation of adherence to prescription will be done at 6 monthly intervals.

ELIGIBILITY:
Inclusion Criteria:

Subjects with IGT in the age group of 30-55 years (n=900) will be identified by screening with a standard OGTT.

Exclusion Criteria:

1. Known diabetes
2. Pregnant women
3. Alcohol abuse
4. Transferable jobs.
5. Subjects with major illness like cancer, hepatic or cardiac diseases.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2014-02 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
1. Rate of conversion of IGT to diabetes. 2. Relative reduction of incidence of diabetes by Sitagliptin among people with IGT compared to Placebo. 3. Increase in reversal of IGT to NGT | At intervals -6 months

SECONDARY OUTCOMES:
1. Beneficial effects in beta cell function. 2. Changes in insulin resistance 3. Improvement in cardiovascular risk factors by Sitagliptin. | Annual

CONTACTS AND LOCATIONS:
Locations (1):
- Dr.Ambady Ramachandran, Chennai, Tamil Nadu, India

REFERENCES:
- [Background] 1.Ramachandran A, Ronald Ma, Snehalatha C. Diabetes in Asia. 2009 Lancet Oct;DOI:10.1016/S0140-6736(09)60937-5. 2.Snehalatha C, Mary S, Selvam S, Sathish Kumar CK, Shetty SB, Nanditha A, Ramachandran A. Changes in insulin secretion and insulin sensitivity in relation to the glycemic outcomes in subjects with impaired glucose tolerance in the Indian Diabetes Prevention Programme-1 (IDPP-1).Diabetes Care. 2009 Oct;32(10):1796-801. 3.Ramachandran A, Snehalatha C, Mary S, Selvam S, Sathish Kumar CK, Catherin Seeli A, Samith Shetty A. Pioglitazone does not enhance effectiveness of life style modification in prevening conversion of impaired glucose tolerance to diabetes in Asian Indians-Results of Indian Diabetes Prevention Programme- (IDPP-2).Diabetologia 2009; 52: 1019 - 1026. 4.Ramachandran A, Snehalatha C. Cardiovascular risk factors in normoglycaemic Asian Indian population-Impact of urbanization. Diabetologia 2009 52; 596-599.